CLINICAL TRIAL: NCT05774002
Title: Psychological Assessment of Scoliosis Patients Undergoing Surgical Management (PASS)
Brief Title: Psychological Assessment of Scoliosis Patients Undergoing Surgical Management
Acronym: PASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-14525
Record Dates: First submitted 2023-02-17; First posted 2023-03-17 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care control groups no psychological intervention (No Intervention): standard of care control groups no psychological intervention
- psychological intervention ADAPT (Experimental): The psychological intervention plan is based on the Aim to Decrease Anxiety and Pain Treatment (ADAPT) model.
  Interventions: Behavioral: Aims to Decrease Anxiety and Pain Treatment (ADAPT)

INTERVENTIONS:
Behavioral: Aims to Decrease Anxiety and Pain Treatment (ADAPT) — One pre-operative and 4 post-operative sessions of cognitive behavioral therapy (CBT) treatment in the first two months, beginning 2-3 weeks after surgery, will be completed.
  Arms: psychological intervention ADAPT

SUMMARY:
Working in partnership with Montefiore-Einstein's Department of Translational Psychiatry, the study team investigators have designed a prospective randomized clinical trial (2:1) study for 45 AIS patients (10-19 yrs.). This protocol includes a baseline assessment of mental health, pain, and function in AIS patients utilizing validated patient reported outcome measures. The investigators will implement and test a structured perioperative psychological intervention program, based on the Aim to Decrease Anxiety and Pain Treatment (ADAPT), which was developed based on evidence-based cognitive behavioral therapy (CBT) protocols for the management of pediatric pain and childhood anxiety disorders

DETAILED DESCRIPTION:
Working in partnership with Montefiore-Einstein's Department of Translational Psychiatry, the investigators have designed a prospective randomized clinical trial (2:1) study for 45 AIS patients (10-19 yrs.). This protocol includes a baseline assessment of mental health, pain, and function in AIS patients utilizing validated patient reported outcome measures. The investigators will implement and test a structured perioperative psychological intervention program, based on the Aim to Decrease Anxiety and Pain Treatment (ADAPT), which was developed based on evidence-based cognitive behavioral therapy (CBT) protocols for the management of pediatric pain and childhood anxiety disorders

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of scoliosis prior to age 20
* Healthy, non-obese aged 10-19 years, with a diagnosis of idiopathic scoliosis, undergoing elective posterior spinal fusion

Exclusion Criteria:

* Diagnosis of scoliosis after age 20
* Permanent cognitive impairment
* Pregnant or breastfeeding women
* Use of opioids in the last 6 months
* Liver or renal diseases and developmental delays

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in Mental health preoperatively and postoperatively using Generalized Anxiety Disorder (GAD-7) | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  Assessing Mental health score changes preoperatively and postoperatively using the Generalized Anxiety Disorder (GAD-7) questionnaire. (GAD-7) questionnaire is a seven-item, self-report anxiety questionnaire. The Scores of 0, 1 or 2 are given for experiencing symptoms 'not at all', for 'several days', for 'more than half the days' and for 'nearly every day', respectively. The scores are then totalled and presented from 0 to 21. Scores of 5, 10 and 15 represent cut-off points for mild, moderate and severe anxiety, respectively. When screening for an anxiety disorder, a recommended cut-off point for referral for further evaluation is 10 or greater.
Assessment of changes in Pain Catastrophizing Scale for Children (PCS-C) preoperatively and postoperatively | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  Pain Catastrophizing Scale for children( PCS-C ) is a 13-item scale One of the main adaptations of the child version of the pain catastrophizing scale is the repetition of the stem "When I have pain, …" at the beginning of each item. Responses for each statement are done using a Likert-type rating scale, ranging from 0 (not at all) to 4 (extremely). A higher score on this scale would indicate a higher level of pain catastrophizing.
Assessment of changes in Mental health preoperatively and post postoperatively using the Patient Health Questionnaire (PHQ)-9. | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders(DSM-IV) criteria as "0" (not at all) to "3" (nearly every day). score of 0-13: no depression. 14-19: mild depression. 20-28: moderate depression. 29-63: severe depression.
Assessment of changes in Mental health preoperatively and postoperatively using PROMIS- (Patient-Reported Outcomes Measurement Information System) short form for Depression | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  PROMIS-short form (Patient-Reported Outcomes Measurement Information System) for Depression is a set of person-centered measures that evaluates mental health in adults and children. PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S.
  PROMIS items consist of a statement (e.g., "I felt alone") with five response options never, rarely, sometimes, often and always.
  PROMIS depression score of less than 50 consider normal. A score of 50= mean of general population sample
Assessment of changes in Mental health preoperatively and postoperatively using PROMIS-(Patient-Reported Outcomes Measurement Information System) v1 short form for Anxiety | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  PROMIS-short form (Patient-Reported Outcomes Measurement Information System) for anxiety is a set of person-centered measures that evaluates mental health in adults and children. PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. PROMIS items consist of a statement (e.g., "I feel fearful") with five response options never, rarely, sometimes, often and always.
  PROMIS anxiety score of less than 50 consider normal. A score of 50= mean of general population reference sample

SECONDARY OUTCOMES:
Assessment of changes in pain preoperatively and postoperatively using Scoliosis Research Society questionnaire-22 revised (SRS-22r) for adolescents with idiopathic scoliosis | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions).
  The pain domain has five questionnaires A score <4 in the SRS-22-r pain domain (1 = severe pain and 5 = pain free) is considered clinically relevant .
Sociodemographic factors using Child Opportunity Index (COI) | preoperatively
  The Child Opportunity Index (COI) 2.0 measures neighborhood resources and conditions that matter for children's healthy development.
  Total represents the overall index, while Education represents the education metrics, Health represents the health & environment metrics, and social & economic represents the social & economic metrics.
  Record sociodemographic factors to assess the impact on treatment adherence and overall outcomes using child opportunity index Child Opportunity Scores are released as metro, state and nationally normed versions. using the nationally normed index conceals within-metro area inequalities because a disproportionate number of neighborhoods are assigned to the "high" and "very high" opportunity levels when referenced to all tracts nationally.
Assessment of changes in mental health preoperatively and postoperatively using Scoliosis Research Society questionnaire-22 revised (SRS-22r) for adolescents with idiopathic scoliosis | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions).
  The mental health domain has five questionnaires:
  5=Best mental health outcome score1=warning score
Assessment of changes in self image score preoperatively and postoperatively using Scoliosis Research Society questionnaire-22 revised (SRS-22r) for adolescents with idiopathic scoliosis | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions).
  The self-image domain has five questionnaires:
  5=Best mental health outcome score1=warning score
Assessment of changes in Function score preoperatively and postoperatively using Scoliosis Research Society questionnaire-22 revised (SRS-22r) for adolescents with idiopathic scoliosis | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions).
  The Function domain has 5 questionnaires:
  5=Best mental health outcome score, 1=warning score
Assessment of changes in Satisfaction with management score preoperatively and postoperatively using Scoliosis Research Society questionnaire-22 revised (SRS-22r) for adolescents with idiopathic scoliosis | preoperatively (baseline), and postoperatively at 6 weeks, 6 months, and 1 year after surgery for both the standard of care control group and psychological intervention group
  The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions).
  The Satisfaction with management domain has 2 questionnaires:
  5=Best mental health outcome score1=warning score
  Are you satisfied with the results of your back management? 5-Very satisfied 4-Satisfied 3-Neither satisfied nor unsatisfied 2-Unsatisfied 1-Very unsatisfied
  Would you have the same management again if you had the same condition? 5-Definitely yes 4-Probably yes 3-Not sure 2-Probably not 1-Definitely not

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Fornari, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marques de Miranda D, da Silva Athanasio B, Sena Oliveira AC, Simoes-E-Silva AC. How is COVID-19 pandemic impacting mental health of children and adolescents? Int J Disaster Risk Reduct. 2020 Dec;51:101845. doi: 10.1016/j.ijdrr.2020.101845. Epub 2020 Sep 10. PMID 32929399
- [Background] Meherali S, Punjani N, Louie-Poon S, Abdul Rahim K, Das JK, Salam RA, Lassi ZS. Mental Health of Children and Adolescents Amidst COVID-19 and Past Pandemics: A Rapid Systematic Review. Int J Environ Res Public Health. 2021 Mar 26;18(7):3432. doi: 10.3390/ijerph18073432. PMID 33810225
- [Background] Raymond C, Provencher J, Bilodeau-Houle A, Leclerc J, Marin MF. A longitudinal investigation of psychological distress in children during COVID-19: the role of socio-emotional vulnerability. Eur J Psychotraumatol. 2022 Jan 24;13(1):2021048. doi: 10.1080/20008198.2021.2021048. eCollection 2022. PMID 35087645
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] Bitsko RH, Claussen AH, Lichstein J, Black LI, Jones SE, Danielson ML, Hoenig JM, Davis Jack SP, Brody DJ, Gyawali S, Maenner MJ, Warner M, Holland KM, Perou R, Crosby AE, Blumberg SJ, Avenevoli S, Kaminski JW, Ghandour RM; Contributor. Mental Health Surveillance Among Children - United States, 2013-2019. MMWR Suppl. 2022 Feb 25;71(2):1-42. doi: 10.15585/mmwr.su7102a1. PMID 35202359
- [Background] Ghandour RM, Sherman LJ, Vladutiu CJ, Ali MM, Lynch SE, Bitsko RH, Blumberg SJ. Prevalence and Treatment of Depression, Anxiety, and Conduct Problems in US Children. J Pediatr. 2019 Mar;206:256-267.e3. doi: 10.1016/j.jpeds.2018.09.021. Epub 2018 Oct 12. PMID 30322701
- [Background] Bitsko RH, Holbrook JR, Ghandour RM, Blumberg SJ, Visser SN, Perou R, Walkup JT. Epidemiology and Impact of Health Care Provider-Diagnosed Anxiety and Depression Among US Children. J Dev Behav Pediatr. 2018 Jun;39(5):395-403. doi: 10.1097/DBP.0000000000000571. PMID 29688990
- [Background] Hutchins HJ, Barry CM, Wanga V, Bacon S, Njai R, Claussen AH, Ghandour RM, Lebrun-Harris LA, Perkins K, Robinson LR. Perceived Racial/Ethnic Discrimination, Physical and Mental Health Conditions in Childhood, and the Relative Role of Other Adverse Experiences. Advers Resil Sci. 2022;3(2):181-194. doi: 10.1007/s42844-022-00063-z. PMID 37181947
- [Background] Zale EL, Lange KL, Fields SA, Ditre JW. The relation between pain-related fear and disability: a meta-analysis. J Pain. 2013 Oct;14(10):1019-30. doi: 10.1016/j.jpain.2013.05.005. Epub 2013 Jul 11. PMID 23850095
- [Background] Page MG, Stinson J, Campbell F, Isaac L, Katz J. Pain-related psychological correlates of pediatric acute post-surgical pain. J Pain Res. 2012;5:547-58. doi: 10.2147/JPR.S36614. Epub 2012 Nov 12. PMID 23204864
- [Background] Rabbitts JA, Groenewald CB, Tai GG, Palermo TM. Presurgical psychosocial predictors of acute postsurgical pain and quality of life in children undergoing major surgery. J Pain. 2015 Mar;16(3):226-34. doi: 10.1016/j.jpain.2014.11.015. Epub 2014 Dec 22. PMID 25540939
- [Background] Batoz H, Semjen F, Bordes-Demolis M, Benard A, Nouette-Gaulain K. Chronic postsurgical pain in children: prevalence and risk factors. A prospective observational study. Br J Anaesth. 2016 Oct;117(4):489-496. doi: 10.1093/bja/aew260. Epub 2016 Oct 17. PMID 28077537
- [Background] Connelly M, Fulmer RD, Prohaska J, Anson L, Dryer L, Thomas V, Ariagno JE, Price N, Schwend R. Predictors of postoperative pain trajectories in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2014 Feb 1;39(3):E174-81. doi: 10.1097/BRS.0000000000000099. PMID 24173016
- [Background] Rabbitts JA, Zhou C, Groenewald CB, Durkin L, Palermo TM. Trajectories of postsurgical pain in children: risk factors and impact of late pain recovery on long-term health outcomes after major surgery. Pain. 2015 Nov;156(11):2383-2389. doi: 10.1097/j.pain.0000000000000281. PMID 26381701
- [Background] Rabbitts JA, Palermo TM, Zhou C, Meyyappan A, Chen L. Psychosocial Predictors of Acute and Chronic Pain in Adolescents Undergoing Major Musculoskeletal Surgery. J Pain. 2020 Nov-Dec;21(11-12):1236-1246. doi: 10.1016/j.jpain.2020.02.004. Epub 2020 Jun 15. PMID 32553622
- [Background] Esteve R, Marquina-Aponte V, Ramirez-Maestre C. Postoperative pain in children: association between anxiety sensitivity, pain catastrophizing, and female caregivers' responses to children's pain. J Pain. 2014 Feb;15(2):157-68.e1. doi: 10.1016/j.jpain.2013.10.007. Epub 2013 Oct 27. PMID 24360639
- [Background] Ramo BA, Collins-Jones TL, Thornberg D, Klinkerman L, Rathjen K, Jo CH. Pain Catastrophizing Influences Preoperative and Postoperative Patient-Reported Outcomes in Adolescent Idiopathic Scoliosis. J Bone Joint Surg Am. 2022 Nov 2;104(21):1859-1868. doi: 10.2106/JBJS.22.00258. Epub 2022 Aug 18. PMID 35984014
- [Background] Rabbitts JA, Fisher E, Rosenbloom BN, Palermo TM. Prevalence and Predictors of Chronic Postsurgical Pain in Children: A Systematic Review and Meta-Analysis. J Pain. 2017 Jun;18(6):605-614. doi: 10.1016/j.jpain.2017.03.007. Epub 2017 Mar 29. PMID 28363861
- [Background] Rabbitts JA, Zhou C, de la Vega R, Aalfs H, Murray CB, Palermo TM. A digital health peri-operative cognitive-behavioral intervention to prevent transition from acute to chronic postsurgical pain in adolescents undergoing spinal fusion (SurgeryPalTM): study protocol for a multisite randomized controlled trial. Trials. 2021 Jul 30;22(1):506. doi: 10.1186/s13063-021-05421-3. PMID 34330321
- [Background] Rabbitts JA, Zhou C, Narayanan A, Palermo TM. Longitudinal and Temporal Associations Between Daily Pain and Sleep Patterns After Major Pediatric Surgery. J Pain. 2017 Jun;18(6):656-663. doi: 10.1016/j.jpain.2017.01.004. Epub 2017 Jan 26. PMID 28131699
- [Background] DiNapoli T.P., Bleiwas K.B., An Economic and Demographic Snapshot of the Bronx. Office of the New York State Comptroller. https://www.osc.state.ny.us/files/reports/osdc/pdf/report-4-2019.pdf
- [Background] Page MG, Campbell F, Isaac L, Stinson J, Katz J. Parental risk factors for the development of pediatric acute and chronic postsurgical pain: a longitudinal study. J Pain Res. 2013 Sep 30;6:727-41. doi: 10.2147/JPR.S51055. eCollection 2013. PMID 24109194
- [Background] Nelson S, Cunningham N. The Impact of Posttraumatic Stress Disorder on Clinical Presentation and Psychosocial Treatment Response in Youth with Functional Abdominal Pain Disorders: An Exploratory Study. Children (Basel). 2020 Jun 2;7(6):56. doi: 10.3390/children7060056. PMID 32498365
- [Background] Cunningham NR, Nelson S, Jagpal A, Moorman E, Farrell M, Pentiuk S, Kashikar-Zuck S. Development of the Aim to Decrease Anxiety and Pain Treatment for Pediatric Functional Abdominal Pain Disorders. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):16-20. doi: 10.1097/MPG.0000000000001714. PMID 28906315
- [Background] Kalomiris AE, Ely SL, Love SC, Mara CA, Cunningham NR. Child-Focused Cognitive Behavioral Therapy for Pediatric Abdominal Pain Disorders Reduces Caregiver Anxiety in Randomized Clinical Trial. J Pain. 2022 May;23(5):810-821. doi: 10.1016/j.jpain.2021.12.001. Epub 2021 Dec 11. PMID 34902549
- [Background] Children's Mental Health: Understanding an Ongoing Public Health Concern, CDC , https://www.cdc.gov/childrensmentalhealth/data.html
- [Background] Dunn J, Henrikson NB, Morrison CC, Blasi PR, Nguyen M, Lin JS. Screening for Adolescent Idiopathic Scoliosis: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Jan 9;319(2):173-187. doi: 10.1001/jama.2017.11669. PMID 29318283
- [Background] Rabbitts JA, Aaron RV, Fisher E, Lang EA, Bridgwater C, Tai GG, Palermo TM. Long-Term Pain and Recovery After Major Pediatric Surgery: A Qualitative Study With Teens, Parents, and Perioperative Care Providers. J Pain. 2017 Jul;18(7):778-786. doi: 10.1016/j.jpain.2017.02.423. Epub 2017 Feb 21. PMID 28232147
- [Background] Davidson F, Snow S, Hayden JA, Chorney J. Psychological interventions in managing postoperative pain in children: a systematic review. Pain. 2016 Sep;157(9):1872-1886. doi: 10.1097/j.pain.0000000000000636. PMID 27355184
- [Background] Sockalingam S, Leung SE, Ma C, Hawa R, Wnuk S, Dash S, Jackson T, Cassin SE. The Impact of Telephone-Based Cognitive Behavioral Therapy on Mental Health Distress and Disordered Eating Among Bariatric Surgery Patients During COVID-19: Preliminary Results from a Multisite Randomized Controlled Trial. Obes Surg. 2022 Jun;32(6):1884-1894. doi: 10.1007/s11695-022-05981-6. Epub 2022 Feb 25. PMID 35218006
- [Background] Charette S, Fiola JL, Charest MC, Villeneuve E, Theroux J, Joncas J, Parent S, Le May S. Guided Imagery for Adolescent Post-spinal Fusion Pain Management: A Pilot Study. Pain Manag Nurs. 2015 Jun;16(3):211-20. doi: 10.1016/j.pmn.2014.06.004. Epub 2014 Nov 6. PMID 25439116
- [Background] Palermo TM, Eccleston C, Lewandowski AS, de C Williams AC, Morley S. Randomized controlled trials of psychological therapies for management of chronic pain in children and adolescents: an updated meta-analytic review. Pain. 2010 Mar;148(3):387-397. doi: 10.1016/j.pain.2009.10.004. Epub 2009 Nov 11. PMID 19910118
- [Background] Vranceanu AM, Barsky A, Ring D. Psychosocial aspects of disabling musculoskeletal pain. J Bone Joint Surg Am. 2009 Aug;91(8):2014-8. doi: 10.2106/JBJS.H.01512. PMID 19651964
- [Background] Vranceanu AM, Bachoura A, Weening A, Vrahas M, Smith RM, Ring D. Psychological factors predict disability and pain intensity after skeletal trauma. J Bone Joint Surg Am. 2014 Feb 5;96(3):e20. doi: 10.2106/JBJS.L.00479. PMID 24500592
- [Background] VanDenKerkhof EG, Peters ML, Bruce J. Chronic pain after surgery: time for standardization? A framework to establish core risk factor and outcome domains for epidemiological studies. Clin J Pain. 2013 Jan;29(1):2-8. doi: 10.1097/AJP.0b013e31824730c2. PMID 23211602
- [Background] Perry M, Starkweather A, Baumbauer K, Young E. Factors Leading to Persistent Postsurgical Pain in Adolescents Undergoing Spinal Fusion: An Integrative Literature Review. J Pediatr Nurs. 2018 Jan-Feb;38:74-80. doi: 10.1016/j.pedn.2017.10.013. Epub 2017 Nov 13. PMID 29167085
- [Background] Basques BA, Bohl DD, Golinvaux NS, Smith BG, Grauer JN. Patient factors are associated with poor short-term outcomes after posterior fusion for adolescent idiopathic scoliosis. Clin Orthop Relat Res. 2015 Jan;473(1):286-94. doi: 10.1007/s11999-014-3911-4. Epub 2014 Sep 9. PMID 25201091
- [Background] Twycross AM, Williams AM, Finley GA. Surgeons' aims and pain assessment strategies when managing paediatric post-operative pain: A qualitative study. J Child Health Care. 2015 Dec;19(4):513-23. doi: 10.1177/1367493514527022. Epub 2014 Apr 11. PMID 24728398
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Weinrib AZ, Azam MA, Birnie KA, Burns LC, Clarke H, Katz J. The psychology of chronic post-surgical pain: new frontiers in risk factor identification, prevention and management. Br J Pain. 2017 Nov;11(4):169-177. doi: 10.1177/2049463717720636. Epub 2017 Jul 12. PMID 29123661
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Parsons B, Schaefer C, Mann R, Sadosky A, Daniel S, Nalamachu S, Stacey BR, Nieshoff EC, Tuchman M, Anschel A. Economic and humanistic burden of post-trauma and post-surgical neuropathic pain among adults in the United States. J Pain Res. 2013 Jun 17;6:459-69. doi: 10.2147/JPR.S44939. Print 2013. PMID 23825931
- [Background] Katz J, Weinrib A, Fashler SR, Katznelzon R, Shah BR, Ladak SS, Jiang J, Li Q, McMillan K, Santa Mina D, Wentlandt K, McRae K, Tamir D, Lyn S, de Perrot M, Rao V, Grant D, Roche-Nagle G, Cleary SP, Hofer SO, Gilbert R, Wijeysundera D, Ritvo P, Janmohamed T, O'Leary G, Clarke H. The Toronto General Hospital Transitional Pain Service: development and implementation of a multidisciplinary program to prevent chronic postsurgical pain. J Pain Res. 2015 Oct 12;8:695-702. doi: 10.2147/JPR.S91924. eCollection 2015. PMID 26508886
- [Background] Katz J, Buis T, Cohen L. Locked out and still knocking: predictors of excessive demands for postoperative intravenous patient-controlled analgesia. Can J Anaesth. 2008 Feb;55(2):88-99. doi: 10.1007/BF03016320. PMID 18245068
- [Background] Goodman JE, McGrath PJ. The epidemiology of pain in children and adolescents: a review. Pain. 1991 Sep;46(3):247-264. doi: 10.1016/0304-3959(91)90108-A. No abstract available. PMID 1758709
- [Background] Voepel-Lewis T, Caird MS, Tait AR, Farley FA, Li Y, Malviya S, Hassett A, Weber M, Currier E, de Sibour T, Clauw DJ. A cluster of high psychological and somatic symptoms in children with idiopathic scoliosis predicts persistent pain and analgesic use 1 year after spine fusion. Paediatr Anaesth. 2018 Oct;28(10):873-880. doi: 10.1111/pan.13467. PMID 30302887
- [Background] Groenewald CB, Law EF, Fisher E, Beals-Erickson SE, Palermo TM. Associations Between Adolescent Chronic Pain and Prescription Opioid Misuse in Adulthood. J Pain. 2019 Jan;20(1):28-37. doi: 10.1016/j.jpain.2018.07.007. Epub 2018 Aug 9. PMID 30098405
- [Background] Harbaugh CM, Lee JS, Hu HM, McCabe SE, Voepel-Lewis T, Englesbe MJ, Brummett CM, Waljee JF. Persistent Opioid Use Among Pediatric Patients After Surgery. Pediatrics. 2018 Jan;141(1):e20172439. doi: 10.1542/peds.2017-2439. Epub 2017 Dec 4. PMID 29203521
- [Background] Perry M. "I thought I was going to die": A meta-synthesis exploring pediatric pain after scoliosis surgery. Int J Orthop Trauma Nurs. 2018 Nov;31:5-12. doi: 10.1016/j.ijotn.2018.09.001. Epub 2018 Sep 6. No abstract available. PMID 30342906
- [Background] LaMontagne LL, Hepworth JT, Cohen F, Salisbury MH. Cognitive-behavioral intervention effects on adolescents' anxiety and pain following spinal fusion surgery. Nurs Res. 2003 May-Jun;52(3):183-90. doi: 10.1097/00006199-200305000-00008. PMID 12792259
- [Background] Johnson JE. Effects of accurate expectations about sensations on the sensory and distress components of pain. J Pers Soc Psychol. 1973 Aug;27(2):261-75. doi: 10.1037/h0034767. No abstract available. PMID 4723974
- [Background] Johnson JE, Fieler VK, Wlasowicz GS, Mitchell ML, Jones LS. The effects of nursing care guided by self-regulation theory on coping with radiation therapy. Oncol Nurs Forum. 1997 Jul;24(6):1041-50. PMID 9243588
- [Background] Powers SW. Empirically supported treatments in pediatric psychology: procedure-related pain. J Pediatr Psychol. 1999 Apr;24(2):131-45. doi: 10.1093/jpepsy/24.2.131. PMID 10361392
- [Background] Kain ZN, Mayes LC, Caramico LA. Preoperative preparation in children: a cross-sectional study. J Clin Anesth. 1996 Sep;8(6):508-14. doi: 10.1016/0952-8180(96)00115-8. PMID 8872693
- [Background] LaMontagne LL. Bolstering personal control in child patients through coping interventions. Pediatr Nurs. 1993 May-Jun;19(3):235-7. PMID 8511003
- [Background] Wall LB, Wright M, Samora J, Bae DS, Steinman S, Goldfarb CA; CoULD Study Group. Social Deprivation and Congenital Upper Extremity Differences-An Assessment Using PROMIS. J Hand Surg Am. 2021 Feb;46(2):114-118. doi: 10.1016/j.jhsa.2020.08.017. Epub 2020 Oct 21. PMID 33097335
- [Background] Chidambaran V, Ding L, Moore DL, Spruance K, Cudilo EM, Pilipenko V, Hossain M, Sturm P, Kashikar-Zuck S, Martin LJ, Sadhasivam S. Predicting the pain continuum after adolescent idiopathic scoliosis surgery: A prospective cohort study. Eur J Pain. 2017 Aug;21(7):1252-1265. doi: 10.1002/ejp.1025. Epub 2017 Mar 27. PMID 28346762
- [Background] Richard HM, Cerza SP, De La Rocha A, Podeszwa DA. Preoperative mental health status is a significant predictor of postoperative outcomes in adolescents treated with hip preservation surgery. J Child Orthop. 2020 Aug 1;14(4):259-265. doi: 10.1302/1863-2548.14.200013. PMID 32874357
- [Background] Richard HM, Nguyen DC, Podeszwa DA, De La Rocha A, Sucato DJ. Perioperative Interdisciplinary Intervention Contributes to Improved Outcomes of Adolescents Treated With Hip Preservation Surgery. J Pediatr Orthop. 2018 May/Jun;38(5):254-259. doi: 10.1097/BPO.0000000000000816. PMID 27328119
- [Background] Baldus C, Bridwell K, Harrast J, Shaffrey C, Ondra S, Lenke L, Schwab F, Mardjetko S, Glassman S, Edwards C 2nd, Lowe T, Horton W, Polly D Jr. The Scoliosis Research Society Health-Related Quality of Life (SRS-30) age-gender normative data: an analysis of 1346 adult subjects unaffected by scoliosis. Spine (Phila Pa 1976). 2011 Jun 15;36(14):1154-62. doi: 10.1097/BRS.0b013e3181fc8f98. PMID 21289576
- [Background] Climent JM, Bago J, Ey A, Perez-Grueso FJ, Izquierdo E. Validity of the Spanish version of the Scoliosis Research Society-22 (SRS-22) Patient Questionnaire. Spine (Phila Pa 1976). 2005 Mar 15;30(6):705-9. doi: 10.1097/01.brs.0000155408.76606.8f. PMID 15770189
- [Background] Carreon LY, Sanders JO, Polly DW, Sucato DJ, Parent S, Roy-Beaudry M, Hopkins J, McClung A, Bratcher KR, Diamond BE; Spinal Deformity Study Group. Spinal appearance questionnaire: factor analysis, scoring, reliability, and validity testing. Spine (Phila Pa 1976). 2011 Aug 15;36(18):E1240-4. doi: 10.1097/BRS.0b013e318204f987. PMID 21343853
- [Background] Pielech M, Ryan M, Logan D, Kaczynski K, White MT, Simons LE. Pain catastrophizing in children with chronic pain and their parents: proposed clinical reference points and reexamination of the Pain Catastrophizing Scale measure. Pain. 2014 Nov;155(11):2360-7. doi: 10.1016/j.pain.2014.08.035. Epub 2014 Aug 29. PMID 25180013
- [Background] Correia, H (2010). PROMIS Statistical Center. Northwestern University. PROMIS Translation Methodology